CLINICAL TRIAL: NCT00182221
Title: A Cohort Study Evaluating the Safety of a Diagnostic Strategy Involving D-Dimer Testing in Patients With Suspected Pulmonary Embolism
Brief Title: Safety of a Diagnostic Strategy With D-Dimer Testing for PE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTMG-2005-SIMPLE; Grant #NA 5154
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Venous Thromboembolism
Keywords: Pulmonary Embolism; Deep Vein Thrombosis; MDA D-Dimer Testing; Diagnostic Algorithm
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: MDA D-Dimer Testing

SUMMARY:
To determine whether D-Dimer testing, using the MDA D-Dimer assay, can be used to simplify the diagnostic process for pulmonary embolism (PE). This will be assessed by performing a cohort study in 1000 patients with suspected PE.

To ascertain if an MDA D-Dimer result of less than 0.75 ug/mL FEU obviates the need for further testing and therapy in patients with suspected PE.

DETAILED DESCRIPTION:
Prospective cohort study of 1000 patients in which those with a negative D-Dimer result undergo no further testing and are followed for 3 months for venous thromboembolism. Patients with a positive D-Dimer undergo standardized testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Suspected PE

Exclusion Criteria:

* Treatment with full-dose anticoagulants for 24 hours or more OR an ongoing requirement for anticoagulants
* Other tests for PE performed prior to eligibility assessment (e.g.other D-Dimer, V/Q scan, pulmonary angiogram, spiral CT, compression ultrasound, venogram).
* Cardiorespiratory instability requiring immediate performance of other tests to diagnose or exclude PE (i.e. inability to wait 30-60 minutes for MDA D-Dimer result)
* Comorbid condition limiting survival to less than three months
* Patient has been asymptomatic for seven days prior to presentation
* Current pregnancy
* Contraindication to contrast (e.g., allergy, renal failure).
* Geographic in accessibility which precludes follow-up
* Presence of central venous catheter (permanent or temporary, including PICC line) at the time of eligibility assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Venousthromboembolism | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Bates, MDCM,MSc, Principal Investigator — Hamilton Health Sciences Corporation
Locations (4):
- Canada (4):
  - St Joseph's Health Care Centre, Hamilton, Ontario
  - Hamilton Health Sciences-Henderson Campus, Hamilton, Ontario
  - Hamilton Health Sciences-McMaster Campus, Hamilton, Ontario
  - Hamilton Health Sciences, General, Hamilton, Ontario